CLINICAL TRIAL: NCT02044120
Title: ESP1/SARC025 Global Collaboration: A Phase I Study of a Combination of the PARP Inhibitor, Niraparib and Temozolomide and/or Irinotecan in Patients With Previously Treated,Incurable Ewing Sarcoma
Brief Title: ESP1/SARC025 Global Collaboration: A Phase I Study of a Combination of the PARP Inhibitor, Niraparib and Temozolomide and/or Irinotecan Patients With Previously Treated, Incurable Ewing Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESP1/SARC025
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Ewing Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing | interventions — niraparib; Temozolomide; Irinotecan

ARMS (3):
- niraparib and temozolomide (Experimental): Niraparib (capsule) and temozolomide (capsule) will be taken together.
  Interventions: Drug: niraparib; Drug: Temozolomide
- niraparib and irinotecan (Experimental): Niraparib will be taken orally and irinotecan will be administered intravenously.
  Interventions: Drug: niraparib; Drug: Irinotecan
- niraparib, irinotecan and temozolomide (Experimental): Niraparib and temozolomide will be taken orally. Irinotecan will be administered intravenously.
  Interventions: Drug: niraparib; Drug: Temozolomide; Drug: Irinotecan

INTERVENTIONS:
Drug: niraparib
Drug: Temozolomide
  Arms: niraparib and temozolomide; niraparib, irinotecan and temozolomide
Drug: Irinotecan
  Arms: niraparib and irinotecan; niraparib, irinotecan and temozolomide

SUMMARY:
The purpose of this study is to define the dose-limiting toxicities and maximum tolerated dose of the poly ADP-ribose polymerase inhibitor niraparib and escalating doses of temozolomide and/or irinotecan in patients with pre-treated incurable Ewing sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Ewing sarcoma
* Evidence of Ewing sarcoma translocation by FISH or RT-PCR.
* Must be willing to undergo tumor biopsy at study entry for biologic correlates.
* If patient > 18 years, must be willing to undergo on-treatment tumor biopsy unless medically contra-indicated
* Recurrent or refractory tumors with no known curative treatment options according to the judgment of the investigator.
* Age ≥ 13 years.
* Life expectancy of ≥ 3 months.
* ECOG performance status 0-2.
* Measurable disease on CT or MRI by RECIST 1.1.
* Adequate organ function
* Patients must have received as a minimum a first line chemotherapy regimen consisting of at least 2 of the following agents: doxorubicin, cyclophosphamide, ifosfamide, etoposide.
* Time elapsed from previous therapy must be ≥ 3 weeks for systemic therapy, ≥ 2 weeks for radiation therapy or major surgery.
* Patients who have undergone autologous hematopoietic stem cell transplantation are eligible once they have recovered from all toxicities from therapy
* Patients who have received allogeneic hematopoietic stem cell transplantation will be eligible 6 months after the procedure provided there is no evidence of active graft-versus-host disease and immunosuppressive treatment has been discontinued for at least 30 days.
* Patients with central nervous system disease are eligible for enrollment if they have received prior radiotherapy or surgery to sites of central nervous system metastatic disease, have been off glucocorticoids for at least 4 weeks, have no overt evidence of neurological deficit and are ≥ 6 weeks from completion of brain irradiation.
* Patients or their legal representative (if the patient is < 18 years old) must be able to read, understand and provide written informed consent to participate in the trial.
* Females of childbearing potential as well as males and their partners must agree to use an effective form of contraception during the study and for 6 months following the last dose of study medication.

Exclusion Criteria:

* Clinically significant unrelated illness which would, in the judgment of the treating physician, compromise the patient's ability to tolerate the investigational agent or be likely to interfere with the study procedures or results.
* Patients with baseline QTc > 480 msec.
* Inability to swallow capsules.
* Known hypersensitivity to any of the components of niraparib or prior hypersensitivity reactions to that class of drugs.
* Known hypersensitivity reaction to temozolomide or any of its components, or dacarbazine (DTIC) if enrolled on ARM 1 or irinotecan or any of its components if enrolled on ARM 2
* Concomitant use of any other investigational or anticancer agent(s).
* Pregnant patients or patients who are breast feeding. Subjects capable of pregnancy (post menarche and not post-menopausal, defined as over 12 months since final menstrual period) must have a negative pregnancy test within 7 days prior to first dose.
* Other clinically significant malignant disease diagnosed within the previous 5 years, excluding intra-epithelial cervical neoplasia or non-melanoma skin cancer.
* Active central nervous system disease.
* Known history of MDS or AML
* Known persistent (> 4 weeks) ≥ Grade 2 neutropenia, ≥ Grade 2 thrombocytopenia or > Grade 3 anemia from prior cancer therapy

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-05; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity and maximum tolerated dose | Approximately 24 months
  Dose limiting toxicity describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment. The maximum tolerated dose is the highest dose of a drug or treatment that does not cause unacceptable side effects.

SECONDARY OUTCOMES:
Tumor response rate | Approximately 24 months
  The percentage of patients whose tumor shrinks or disappears after treatment
Progression-free survival | Month 4 and 6
  The time from starting treatment until disease progression
Duration of response | Approximately 24 months
  The time from tumor response to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Chugh, MD, Principal Investigator — University of Michigan; Sandra Strauss, MBBS, PhD, Principal Investigator — University College London, Cancer Institute
Locations (5):
- United States (4):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - National Cancer Institute, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Seattle's Children Cancer Center, Seattle, Washington
- University College London Hospital, London, United Kingdom

REFERENCES:
- [Derived] Chugh R, Ballman KV, Helman LJ, Patel S, Whelan JS, Widemann B, Lu Y, Hawkins DS, Mascarenhas L, Glod JW, Ji J, Zhang Y, Reinke D, Strauss SJ. SARC025 arms 1 and 2: A phase 1 study of the poly(ADP-ribose) polymerase inhibitor niraparib with temozolomide or irinotecan in patients with advanced Ewing sarcoma. Cancer. 2021 Apr 15;127(8):1301-1310. doi: 10.1002/cncr.33349. Epub 2020 Dec 8. PMID 33289920